CLINICAL TRIAL: NCT04577274
Title: Impact of High Protein and Low Carbohydrate Smoothie Drinks Versus Diabetes-specific Nutritional Formulas on Postprandial Glucose Homeostasis in Type-2 Diabetes Mellitus
Brief Title: Impact of High Protein and Low Carbohydrate Smoothie Drinks in Type-2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 814/2562 (IRB3)
Record Dates: First submitted 2020-10-01; First posted 2020-10-06 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: clinical nutrition; smoothie drink; meal replacement; medical food; diabetes; obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Obesity | interventions — Glucerna

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- smoothie with regular formulas (SM) (Experimental): Participants were given 300 kcal smoothie with regular formulas within 3-5 minutes and blood collection after drinking at 30, 60, 90, 120, 180 and 240 minutes.
  Interventions: Dietary Supplement: smoothie with regular formulas (SM)
- smoothie with low carbohydrate formulas (SMLS) (Experimental): Participants were given 300 kcal smoothie with low carbohydrate formulas within 3-5 minutes and blood collection after drinking at 30, 60, 90, 120, 180 and 240 minutes.
  Interventions: Dietary Supplement: smoothie with low carbohydrate formulas (SMLS)
- conventional diabetic enteral drinks (Glucerna) (Active Comparator): Participants were given 300 kcal Glucerna within 3-5 minutes and blood collection after drinking at 30, 60, 90, 120, 180 and 240 minutes.
  Interventions: Dietary Supplement: conventional diabetic enteral drinks (Glucerna)

INTERVENTIONS:
Dietary Supplement: smoothie with regular formulas (SM) — Participants were given 300 kcal of smoothie drink within 3-5 minutes and blood collection after drinking at 30, 60, 90, 120, 180 and 240 minutes. Participants have one week wash out period before try-out other formulas.
  Arms: smoothie with regular formulas (SM)
Dietary Supplement: smoothie with low carbohydrate formulas (SMLS) — Participants were given 300 kcal of smoothie drink within 3-5 minutes and blood collection after drinking at 30, 60, 90, 120, 180 and 240 minutes. Participants have one week wash out period before try-out other formulas.
  Arms: smoothie with low carbohydrate formulas (SMLS)
Dietary Supplement: conventional diabetic enteral drinks (Glucerna) — Participants were given 300 kcal of smoothie drink within 3-5 minutes and blood collection after drinking at 30, 60, 90, 120, 180 and 240 minutes. Participants have one week wash out period before try-out other formulas.
  Arms: conventional diabetic enteral drinks (Glucerna)

SUMMARY:
We compared between a regular high protein or a high protein and low carbohydrate smoothie drinks with conventional diabetic enteral drinks (Glucerna) on glucose homeostasis, insulin and lipid metabolism in type 2 diabetic and obese individuals.

DETAILED DESCRIPTION:
We aimed to determine the effect of high protein and low carbohydrate smoothie drinks on glucose homeostasis, insulin and lipid metabolism in type 2 diabetic and obese individuals. We compared between a regular high protein or a high protein and low carbohydrate smoothie drinks with conventional diabetic enteral drinks (Glucerna). A crossover design study was done in 60 diabetic participants. Participants consumed 300 kilocalories of each drink at a time with one week wash out period between drinks and glucose response curves at baseline, 30, 60, 90, 120, 180 and 240 minutes were monitored and compared. The products were formulated to supply 1 kilocalorie/milliliter (kcal/ml). Dietary compositions in regular formulas (smoothie, SM) were 30-40% carbohydrate, 20-30% protein and 30-50% fat. While in smoothie with low carbohydrate formulas (SMLS), they were 25-35% carbohydrate, 25-30% protein and 35-55% fat vs. a control formula (Glucerna).

ELIGIBILITY:
Inclusion Criteria:

1. people with type 2 diabetes mellitus or use blood glucose-lowering drugs more than 3 months
2. BMI > 25 kg/m^2
3. HbA1c 6.5 - 8.5
4. use stable level of blood glucose-lowering drugs and blood lipid-lowering drugs more than 3 months

Exclusion Criteria:

1. pregnancy or breastfeeding
2. people with chronic diseases or tube feeding or dysphagia i.e. pneumonia
3. people with insulin injection or use GLP-1 analogues drugs or DPP-4 inhibitors drugs
4. people with history of bariatric surgery, gastroparesis, malabsorption
5. people with history of diseases that affect blood glucose/lipid control i.e. hyperthyroidism, endocrinology and kidney disorders
6. use long-term immunosuppressants
7. cancer patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Glycemia at 240 minutes | Minutes after intake of each smoothie formula: 0, 30, 60, 90, 120, 180, 240
  glucose (mg/dl)
Change from baseline Insulin at 240 minutes | Minutes after intake of each smoothie formula: 0, 30, 60, 90, 120, 180, 240
  insulin (μU/ml)

SECONDARY OUTCOMES:
Age | Baseline
  years
Weight | Baseline
  kg
Height | Baseline
  cm
Body Mass Index | Baseline
  kg/m^2
Waist circumference | Baseline
  cm
Blood pressure | Baseline
  Systolic and Diastolic blood pressure (mmHg)
Complete Blood Count (CBC) | Baseline
  Red blood cells (RBC) [10^6 cells/ul], White blood cells (WBC) [10^3 cells/ul], Hemoglobin (HGB) [g/dL], Hematocrit (HCT) [%]
glycosylated hemoglobin (HbA1C) | Baseline
  percentage (%)
liver aminotransferaces activity - Serum glutamate oxaloacetate transaminase (SGOT) | Baseline
  Serum glutamate oxaloacetate transaminase (SGOT) [U/L]
liver aminotransferaces activity - Serum glutamate pyruvate transaminase (SGPT) | Baseline
  Serum glutamate pyruvate transaminase (SGPT) [U/L]
lipid profiles concentration analysis | Baseline
  Triglycerides (mg/dl), Cholesterol (mg/dl), HDL-Cholesterol (mg/dl) and LDL-Cholesterol (mg/dl)
Creatinine concentration analysis | Baseline
  mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Korapat Mayurasakorn, MD., Principal Investigator — Doctor in Family Medicine
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand